CLINICAL TRIAL: NCT00761124
Title: Informed Decision-Making Regarding PSA Screening
Brief Title: Informed Decision-Making Regarding Prostate Specific Antigen (PSA) Screening in 50-70 Year Old Latino Men
Acronym: PSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-001693; R01CA102486 (NIH)
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: PSA screening; Prostate cancer and Latino men
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Educational small group session regarding prostate cancer
  Interventions: Behavioral: Intervention Session
- 2 (Other): Printed material regarding general prostate cancer information provided.
  Interventions: Behavioral: Printed Material

INTERVENTIONS:
Behavioral: Intervention Session — A one-hour discussion group composed of 8-10 Latino men. The session includes an interactive, multimedia presentation led by a facilitator to guide participant interaction.
  Arms: 1
Behavioral: Printed Material — General prostate cancer pamphlet
  Arms: 2

SUMMARY:
The purpose of this intervention trial is aiming to increase inform decision- making in Latino men regarding prostate cancer screening.

The investigators propose to find out how much Latino men know about the benefits and risks of prostate cancer screening and what factors influence how they decide whether or not to have screening. The investigators are also interested in learning how providing education information, both verbally and in print, about the risks and benefits of prostate cancer screening affects men's interest and knowledge.

The intervention is an interactive multi-media presentation made up of a small group of 8-10 Latino men gathered to discuss about prostate cancer, screening methods, treatment, and the controversy within the medical community regarding PSA screening. A facilitator guides the 1-hour discussion and encourages participant interaction. The effect of this intervention was tested on 1000 Latino men within Los Angeles county.

Participants were recruited from 38 community venues (churches, community center, etc.). All participants were interviewed before being randomized to receive written (control group) or oral (intervention) prostate cancer education material. All of the participants will be followed up at 6-months via a telephone interview.

The investigators hypothesize that the intervention group will have an increase knowledge of prostate cancer, will have increase communication with family, friends, and medical provider, and will have an increase rate of PSA screening compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Latino men
* 50 to 70 years old
* Not ever having prostate biopsy
* Not ever having prostate cancer
* Not having had a PSA test within the past 12 months
* Not having BPH (prostate inflammation)
* Not currently experiencing prostate problems such as pain or burning sensation during urination, blood in urine, and/or desire to urinate frequently

Exclusion Criteria:

* Not Latino
* Younger than 50 or older than 70 years old
* Currently experiencing prostate problems such as pain or burning sensations while urinating, blood in urine, and/or desire to urinate frequently
* Living outside of Los Angeles county
* Having had a prostate biopsy
* Having had prostate cancer previously
* Having had a prostatectomy

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2003-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Inform Decision-Making | 6 months post-baseline interview

SECONDARY OUTCOMES:
Prostate cancer knowledge, Receipt of PSA, and Communication with family, friends, and medical providers | 6 months post-baseline interview

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Division of Cancer Prevention and Control Research, Los Angeles, California, United States